CLINICAL TRIAL: NCT06918080
Title: Hepatoprotective Measures for Children at High Risk of Non Alcoholic Fatty Liver Disease
Brief Title: Hepatoprotective Measures for Children at High Risk of NAFLD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU MD300/2023; FMASU MD300/2023 (Other: Faculty on Medicine Ain Shams University Research Ethical Committee)
Record Dates: First submitted 2025-01-07; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Non Alcoholic Fatty Liver Diseases (NAFLD); Obesity and Overweight; Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Obesity; NAFLD
MeSH Terms: conditions — Obesity; Overweight; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Non-alcoholic Fatty Liver Disease | interventions — Ursodeoxycholic Acid; Docosahexaenoic Acids; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm (1) (Experimental): Patients will follow Mediterranean Diet (MD) for 12 weeks, this diet is characterized by a high intake of vegetables, fruit, whole cereals, legumes, nuts, and fish and a low intake of red meat and homemade desserts. The main added fat is extra virgin olive oil, with 35-40% kcal from fat (<10% from saturated fat), 40-44% kcal from carbohydrate, and 20% kcal from protein. Patient caloric intake will be calculated according to the Recommended Daily Allowance (RDA) for age.
  Supplementation of omega 3, the dose of omega-3 fatty acids will be determined by baseline weight (<40 kg-450 mg/day, 40-60 kg-900 mg/day, >60 kg-1300 mg/day).
  Patients will also receive daily doses of Ursodeoxycholic acid (UCD) Ursofalk) in a dose of 20 mg/Kg/day in two divided doses depending on their body weight for 12 weeks. Patients will participate in a 12-week exercise program for 30-45 min/day for 3 days/week in the first 2 weeks and for 60 min/day for 4-5 days/week thereafter.
  Interventions: Drug: Ursodeoxycholic Acid 250 Mg Oral Capsule; Dietary Supplement: Omega -3 fatty acids; Behavioral: Physical exercise; Behavioral: Mediterrenean diet
- Arm(2) (Active Comparator): Patients will receive lifestyle modification according to NASPGHAN Clinical Guidelines for the treatment of NAFLD in Children. Patients will follow healthy and well-balanced diet. Patient caloric intake will be calculated according to the Recommended Daily Allowance (RDA) for age with avoidance of sugar-sweetened beverages, moderate- to high-intensity exercise daily will be encouraged, and screen time will be limited to less than 2 hours.
  Interventions: Behavioral: Diet according to NASPGHAN guidelines

INTERVENTIONS:
Drug: Ursodeoxycholic Acid 250 Mg Oral Capsule — Daily doses of Ursodeoxycholic acid (UCD) Ursofalk) in a dose of 20 mg/Kg/day in two divided doses depending on their body weight for 12 weeks will be assigned to arm(1)
  Arms: Arm (1)
Dietary Supplement: Omega -3 fatty acids — Supplementation of omega 3, the dose of omega-3 fatty acids will be determined by baseline weight (<40 kg-450 mg/day, 40-60 kg-900 mg/day, >60 kg-1300 mg/day) will be assigned to children in arm (1). Side effect such as gastrointestinal upset and allergy will be monitored, compliance will be monitored by weekly phone call
  Arms: Arm (1)
Behavioral: Physical exercise — Patients assigned to arm (1) will participate in a 12-week exercise program for 30-45 min/day for 3 days/week. in the first two weeks and for 60 min/day for 4-5 days/week in the following weeks
  Arms: Arm (1)
Behavioral: Mediterrenean diet — Patients in arm (1) will follow Mediterranean Diet (MD) for 12 weeks, this diet is characterized by a high intake of vegetables, fruit, whole cereals, legumes, nuts, and fish and a low intake of red meat and homemade desserts. The main added fat is extra virgin olive oil, with 35-40% kcal from fat (<10% from saturated fat), 40-44% kcal from carbohydrate, and 20% kcal from protein.( Plaz et al., 2019) Patient caloric intake will be calculated according to the Recommended Daily Allowance (RDA) for age.
  Compliance to the MD will be assessed in all patients using the KIDMED index at 4 ,8 and 12 weeks.Those who prove to be non-compliant will be excluded from the study.
  Arms: Arm (1)
Behavioral: Diet according to NASPGHAN guidelines — Patients in arm (2) will receive lifestyle modification according to NASPGHAN Clinical Guidelines for the treatment of NAFLD in Children. Patients will follow healthy and well-balanced diet. Patient caloric intake will be calculated according to the Recommended Daily Allowance (RDA) for age, with avoidance of sugar-sweetened beverages, moderate- to high-intensity exercise daily will be encouraged, and screen time will be limited to less than 2 hours.
  Arms: Arm(2)

SUMMARY:
Non Alcoholic Fatty Liver Disease (NAFLD) is a spectrum of disease, ranging from simple fatty deposition (steatosis) to inflammation (steatohepatitis), fibrosis, cirrhosis, and end-stage liver failure. In childhood, it may be associated with a metabolic syndrome or with obesity, or even in normal children. Liver biopsy has always been the gold standard method for diagnosing and staging NAFLD. However, the urge of non-invasive biomarkers or imaging techniques has been recommended. This study will evaluate the use of the LIVERFASt biomarkers for early detection and staging of NAFLD.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD), defined as abnormal hepatic accumulation of macrovesicular fat in the absence of other etiologies. NAFLD is becoming increasingly prevalent in the pediatric population in direct correlation with the emergence of childhood obesity as a significant pediatric health problem.

Most patients with NAFLD are asymptomatic, and the disease is detected incidentally. Some patients complain of fatigue, malaise, and vague right upper abdominal discomfort. The most common signs are hepatomegaly and laboratory abnormalities, which include a 2 to 4 fold elevation of serum aminotransferase levels, while other liver function test results are usually normal unless advanced liver disease is present. Most are obese, many have diabetes mellitus, hypercholesterolemia, or hypertriglyceridemia.

This study will recruit 195 children aged between 5-18 years divided in 3 groups, each 65 participants: (P1) overweighted (BMI between 84th& 94 th centiles) or obese (BMI>95th)and (P2) children on maintenance chemotherapy for acute lymphoblastic leukemia at risk for NAFLD, compared with control healthy children matched for gender and age (P3). Each participant will be subjected to history taking , clinical examination and anthropometric measures: weight,height,BMI,waist circumference and triceps skin fold thickness. Body composition will also be done.

Thereafter each participant will have a baseline LIVERFASt, U/S and Transient elastography assessments and will be randomly assigned by a computer based program to one of two interventional arms: Arm(1): which comprises Mediterranean Diet (MD) for 12 weeks, Supplementation of omega 3, the dose of omega-3 fatty acids will be determined by baseline weight (<40 kg-450 mg/day, 40-60 kg-900 mg/day, >60 kg-1300 mg/day), daily doses of Ursodeoxycholic acid (UCD)( Ursofalk) in a dose of 20 mg/Kg/day in two divided doses depending on their body weight for 12 weeks and a 12-week exercise program for 30-45 min/day for 3 days/week. in the first two weeks and for 60 min/day for 4-5 days/week in the following weeks. In Arm(2), Patients will receive lifestyle modification according to NASPGHAN Clinical Guidelines for the treatment of NAFLD in Children. Patients will follow healthy and well-balanced diet. Patient caloric intake will be calculated according to the Recommended Daily Allowance (RDA) for age ) with avoidance of sugar-sweetened beverages, moderate- to high-intensity exercise daily will be encouraged, and screen time will be limited to less than 2 hours. The group of patients on chemothrapy will all receive arm(1) intervention without randomization,so as not to deprive them from the hypothecal benefit of the intervention.

LIVERFASt evaluation and imaging will be repeated by the end of the 12 week intervention period as follow up

Screening for NAFLD is appropriate because it can be detected before the onset of irreversible, end-stage liver disease. Identification of children with NAFLD is important because effective treatment is available. Although more challenging to implement than prescribing a medication, lifestyle intervention can be effective at reversing NAFLD and even NASH, particularly if initiated early in the course of disease, before advanced fibrosis has developed.

Although liver biopsy is the current standard to provide critical diagnostic and staging information, including the presence of NASH, and to eliminate alternative and/or concurrent diagnoses. Liver biopsy has inherent limitations for staging NAFLD because of the non uniformity of disease throughout the liver in reference to the small sample of liver obtained Other noninvasive methods used as screening tests for NAFLD include measurement of liver stiffness through transient elastography, which is an accurate and reproducible methodology to identify pediatric subjects without fibrosis or significant fibrosis, or with advanced fibrosis.

LIVERFASt (LF)is a panel of three non-invasive patented artificial intelligence neural networks algorithms estimating liver fibrosis (LF-Fib), inflammatory activity (LF-Act) and steatosis (LF-Ste) intended for the evaluation of NAFLD risk patients. It combines age, gender and BMI with ten serum biomarkers easy to determine in routine biochemistry in fasting patients that are independently correlated with the severity of each histological feature of nonalcoholic fatty liver disease (NAFLD).

This study evaluates the use of the LIVERFASt biomarkers as well as ultrasound (US) for early detection and staging of NAFLD, and the impact of a designed non-invasive therapeutic intervention in the form of Omega-3, Ursodeoxycholic acid and lifestyle modification, in 2 groups of children compared with a control group of healthy children age and gender matched.

ELIGIBILITY:
Inclusion Criteria:

Children aged between 5-18 years, including:

* Population P1: N=65 overweight (BMI between 85th & 94th centile) and obese children (BMI = or > 95th centile) at-risk of NAFLD
* Population P2: N=65 children on maintenance therapy (High Dose Methotrexate 2.5 or 5 mg according to risk level, every other week for 4 doses and daily 6-Mercaptopurine tab. 50 mg/m2/day for 56 days) for Acute Lymphoblastic Leukemia, at risk of chemotherapy induced steatohepatitis.
* Population P3: N=65 control healthy children matched for gender and age with P1&2.

Exclusion Criteria:

* Conditions that could interfere with measured labs (acute/chronic hemolysis, acute hepatitis, extra hepatic cholestasis, systemic inflammatory response).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Study of the prevalence of liver steatosis, steatohepatitis and fibrosis among the study population by using LIVERFASt. | 2 years
  Study of the prevalence of liver steatosis, steatohepatitis and fibrosis among the study population by using LIVERFASt.

SECONDARY OUTCOMES:
To compare the prevalence of NAFLD as estimated by LIVERFASt ,in two paediatric populations: who use chemotherapy for hematologic malignancies, and other who are at high risk of NAFLD(obese and overweighted)with apparently healthy controls matched for ge | 2 years
  To compare the prevalence of NAFLD as estimated by LIVERFASt ,in two paediatric populations: who use chemotherapy for hematologic malignancies, and other who are at high risk of NAFLD(obese and overweighted)with apparently healthy controls matched for gender and age.

OTHER OUTCOMES:
To estimate the efficacy and safety of therapeutic interventions in the form of Omega-3 supplements, Ursodeoxycolic acid and life style changes by assessment of the side effects, and their efficacy on liver fibrosis, steatosis and steatohepatitis. | 2 years
  To estimate the efficacy and safety of therapeutic interventions in the form of Omega-3 supplements, Ursodeoxycolic acid and life style changes by assessment of the side effects, and their efficacy on liver fibrosis, steatosis and steatohepatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Manal H El-Sayed, Professor of pediatrics, Principal Investigator — Ain Shams University-Faculty of Medicine-Pediatric Department; Fatma SE Ebeid, Professor of pediatrics, Study Chair — Ain Shams University-Faculty of Medicine-Pediatric Department
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo
  - Faculty of Medicine Ain Shams Research Institute- Clinical Research Center (MASRI-CRC), Cairo

IPD SHARING:
Plan to Share IPD: Undecided
For the sake of patients' confidentiality and dignity